CLINICAL TRIAL: NCT07248670
Title: Concurrent Chemoradiotherapy With or Without Metronomic Capecitabine in High-Risk T1-2N1M0 Nasopharyngeal Carcinoma: A Multicenter, Randomized Controlled, Phase III Clinical Study
Brief Title: Concurrent Chemoradiotherapy With or Without Metronomic Capecitabine in High-Risk T1-2N1M0 NPC
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Chongqing University Cancer Hospital (Other)
Responsible Party: Principal Investigator, Ying Wang, Director of the hospital, Chongqing University Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CZLL2025-031-001
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Nasopharyngeal Cancinoma (NPC)
Keywords: Nasopharyngeal Carcinoma; Metronomic Capecitabine; EBV DNA
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Capecitabine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- observation (No Intervention): observation after CCRT
- metronomic adjuvant chemotherapy with capecitabine (Experimental): metronomic adjuvant chemotherapy with capecitabine after CCRT.
  Interventions: Drug: metronomic adjuvant chemotherapy with capecitabine

INTERVENTIONS:
Drug: metronomic adjuvant chemotherapy with capecitabine — The concurrent chemoradiotherapy (CCRT) regimen consisted of IMRT delivering 69.96 Gy in 33 fractions, combined with cisplatin administered at 35-40 mg/m² weekly for 6 cycles to achieve a cumulative dose of ≥200 mg/m².
  During CCRT, plasma EBV DNA titer was monitored weekly. If EBV DNA remained undetectable from the second week after CCRT initiation until the end of radiotherapy, patients underwent observation after radiotherapy. If EBV DNA was detectable at any time point from the second week of CCRT until the end of radiotherapy, patients were randomized in a 1:1 ratio to observation or metronomic adjuvant chemotherapy with capecitabine (650 mg/m² twice daily, Q3W) for 8 cycles (6 months) after radiotherapy.
  Arms: metronomic adjuvant chemotherapy with capecitabine

SUMMARY:
This Phase III multicenter trial investigates treatment intensification for high-risk, stage T1-2N1M0 nasopharyngeal carcinoma. Patients with high-risk features (>3 metastatic lymph nodes, necrosis, or confluence) receive concurrent chemoradiotherapy. Those with detectable EBV DNA during radiotherapy are randomized 1:1 to adjuvant capecitabine or observation alone to assess efficacy and safety

DETAILED DESCRIPTION:
This is a multicenter, randomized, phase III trial enrolling patients with AJCC/UICC 9th edition stage T1-2N1M0 nasopharyngeal carcinoma who have at least one of the following high-risk features: more than 3 metastatic cervical lymph nodes, presence of nodal necrosis, or presence of nodal confluence. All patients receive concurrent chemoradiotherapy (CCRT) with a weekly cisplatin regimen. Plasma EBV DNA is monitored weekly during CCRT. High-risk patients with detectable EBV DNA at any time from the second week of CCRT until the end of radiotherapy are randomized in a 1:1 ratio to receive either metronomic adjuvant chemotherapy with capecitabine or follow-up observation alone, to evaluate the efficacy and safety of treatment intensification

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 70 years.
2. Pathologically confirmed, previously untreated "non-keratinizing carcinoma (WHO types II/III)" of the nasopharynx.
3. Diagnosed as stage T1-2N1M0 (Stage IB) according to the 9th edition of the American Joint Committee on Cancer/Union for International Cancer Control (AJCC/UICC) staging system.
4. Presence of at least one of the following high-risk lymph node features: more than three metastatic cervical lymph nodes (retropharyngeal lymph nodes are not counted), presence of nodal necrosis, or presence of nodal confluence.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. Detectable baseline plasma EBV DNA, with EBV DNA remaining detectable at any time point from the second week after the start of concurrent chemoradiotherapy until the end of radiotherapy.
7. Adequate bone marrow function, liver and renal function.

Exclusion Criteria:

1. Intolerance or allergy to capecitabine.
2. Conditions that may interfere with the absorption or adherence to oral medication, such as dysphagia, chronic diarrhea, or intestinal obstruction.
3. Administration of biologic therapy or immunotherapy during or prior to radiotherapy.
4. Pregnancy or lactation (a pregnancy test should be considered for women of childbearing potential, and emphasis must be placed on effective contraception during the treatment period).
5. Any concurrent severe or uncontrolled medical condition that would pose an unacceptable risk or compromise protocol compliance, including but not limited to untreated unstable cardiac disease, renal disease, chronic hepatitis, poorly controlled diabetes (fasting blood glucose >1.5×ULN), or mood disorders.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2025-10-04 (Actual); Primary Completion 2031-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
FFS | 3-year
  FFS is defined as the time from randomization to the first occurrence of local regional recurrence, distant metastasis, or death from any cause

SECONDARY OUTCOMES:
DMFS | 3-year
LRRFS | 3-year
OS | 3-year

CONTACTS AND LOCATIONS:
Locations (1):
- Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
Due to ethical considerations, contact us via email if needed.